CLINICAL TRIAL: NCT05662488
Title: 68Ga-FAPI PET for Response Evaluation and Prognosis Prediction in Advanced Liver and Biliary Cancer Patients Treated With PD-1 Based Combination Therapy: A Head-to-head Comparison to 18F-FDG PET
Brief Title: FAPI PET for Response Evaluation and Prognosis Prediction in Liver and Biliary Cancer Patients Treated With PD-1 Combination Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-FAPI-LBC-RESPONSE
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma; Bile Duct Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: [68Ga]FAPI PET/CT and [18F]FDG PET/CT — To perform [68Ga]FAPI PET/CT and [18F]FDG PET/CT in patients with advanced liver and biliary cancer before and after treatment with PD-1 Based Combination Therapy

SUMMARY:
The purpose of this study is to explore the ability of positron emission tomography (PET) with [68Ga]FAPI to detect, evaluate treatment response, and predict prognosis in advanced liver and biliary cancer patients treated with anti-PD-1 antibodies-based combination therapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) and bile tract cancers (BTC) are major health issue worldwide, particularly in Eastern Asia. Anti-PD-1 antibodies-based combination therapy has shown considerable efficacy in advanced HCC and BTC. However, an objective response is only achieved in a portion of patients. Thus, there is an urgent need for better patient selection before immunotherapy as well as accurate evaluation of treatment response.

PET is a noninvasive imaging technique which might be an effective tool for evaluating anti-PD-1 antibody-based combination treatment in liver and biliary cancer. 68Ga-FAPI has been developed as a novel agent targeting fibroblast activation protein (FAP) that is overexpressed in cancer-associated fibroblasts in liver and biliary cancer. Prior studies have shown that FAP-expressing CAF suppresses anti-tumor immunity while suppressing FAP can overcome stromal barriers to immuno-oncological responses. Meanwhile, 68Ga-FAPI PET showed a high detection rate in primary and metastatic lesions in liver and biliary cancer. The aim of this study is to evaluate the ability of positron emission tomography (PET) with [68Ga]FAPI to detect, evaluate treatment response, and predict prognosis in advanced liver and biliary cancer patients treated with anti-PD-1 antibodies-based combination therapy. Our hypothesis is that baseline [68Ga]FAPI PET parameters can predict response and clinical benefit of anti-PD-1 antibodies-based combination therapy and overall survival; that effects of anti-PD-1 antibodies-based combination therapy in liver and biliary cancer can be detected and quantified by [68Ga]FAPI PET after treatment in correlation with other radiological findings and clinical endpoints; that such effects are more prominent with [68Ga]FAPI PET than with the traditional [18F]FDG PET.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic and/or unresectable HCC or BTC
* Child Pugh A or B liver function status
* an ECOG performance status score of 0-2

Exclusion Criteria:

* intolerance to anti-PD-1-based combination therapy
* active or prior autoimmune disease
* concurrent use of immunosuppressive medicaments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced HCC or BTC patients who accept PD1-based combination therapy
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Baseline SUVmax on [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 2 years
  Baseline FAPI and FDG SUVmax, fibro-activation tumor volume (metabolic tumor volume), total lesion fibro-activation (total lesion glycolysis) before treatment were determined.
Baseline active tumor volume on [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 2 years
  Baseline fibro-activation tumor volume and metabolic tumor volume before treatment were determined.
Baseline total lesion activation on [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 2 years
  Baseline total lesion fibro-activation and total lesion glycolysis before treatment were determined.
Response of SUVmax to anti-PD1-based combination therapy shown in [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 1 years
  Changes in FAPI and FDG SUVmax during treatment were determined.
Response of active tumor volume to anti-PD1-based combination therapy shown in [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 1 years
  Changes in fibro-activation tumor volume and metabolic tumor volume during treatment were determined.
Response of total lesion activation to anti-PD1-based combination therapy shown in [68Ga]FAPI and [18F] FDG PET Scans | through study completion, an average of 1 years
  Changes in total lesion fibro-activation and total lesion glycolysis during treatment were determined.

SECONDARY OUTCOMES:
Tumor response evaluated by CT and MRI | through study completion, an average of 1 years
  Tumor response was reported per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
Overall survival after treatment | through study completion, an average of 2 years
  Overall survival after treatment
Progression-free survival after treatment | through study completion, an average of 2 years
  Progression-free survival after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Beijing, China